CLINICAL TRIAL: NCT06230718
Title: Upper Limb Electromyographic Response to Motor Imagery and Action Observation in Acquired Brain Injury Patients.
Brief Title: EMG Analysis in ABI: Motor Imagery and Action
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Ana María Martín Nogueras, Principal Investigator, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIAO
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Quality of Life; Mirror Movement
Keywords: Stroke rehabilitation; Electromyography; Neuroplasticity; Upper Linb; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Masking Description: Patients will receive 3 interventions: placebo, motor imagery and action observation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): The intervention group will receive 3 experimental procedures
  1. Placebo control
  2. Motor Imagery- Active Comparator
  3. Action Observation (OA) Active comparator muscle activation control by surface electromyography will be recorded in these three situations
  Interventions: Other: Motor Imagery (MI); Other: Action Observation (AO); Other: Control condition- placebo

INTERVENTIONS:
Other: Motor Imagery (MI) — mental process where an individual visualizes or imagines themselves performing a movement without actually executing it physically. This cognitive process involves the mental rehearsal of motor actions, engaging similar neural pathways that are used when physically performing the action.
Other: Action Observation (AO) — rehabilitation technique based on the principle of observing actions to improve motor function and learning. This approach is rooted in the concept of the mirror neuron system, a group of neurons that are activated both when a person performs an action and when they observe the same action performed by others.
Other: Control condition- placebo — Recording with images of landscapes without the presence of any person or animal that could evoke MI or OA.

SUMMARY:
This study focuses on electromyographic analysis of upper limb muscle activation in stroke survivors during Motor Imagery (MI) and Action Observation (AO) rehabilitation techniques. By measuring muscle activity in the wrist and finger flexors and extensors, the research seeks to understand the impact of MI and AO on motor function recovery post-stroke. Conducted at the University of Salamanca, the study involves stroke survivors participating in a series of three experimental sessions. The analysis will correlate electromyographic responses with functional independence, limb functionality, and cognitive factors. The research aims to contribute to the fields of occupational therapy and physiotherapy, offering insights into effective rehabilitation methods for improving quality of life in stroke survivors.

DETAILED DESCRIPTION:
This study investigates muscle activation in the upper limbs of stroke survivors using electromyographic analysis during Motor Imagery (MI) and Action Observation (AO). Stroke, a major cause of disability, often results in motor impairments in the upper limb, impacting daily activities. The research focuses on innovative rehabilitation techniques based on neuroplasticity, such as MI and AO, stimulated by the discovery of mirror neurons.

The primary goal is to record upper limb muscle activation during MI and AO, using surface electromyography to measure activation in wrist and finger flexors and extensors. The study will also explore the relationship between electromyographic responses and factors like daily activity independence, limb functionality, quality of life, mental evocation ability, and cognitive impairment.

Conducted at the University of Salamanca, the study will recruit stroke survivors for a three-session experimental protocol involving control, MI, and AO conditions. Data will be analyzed with SPSS Statistics, ensuring anonymity and ethical compliance. The research aims to enhance understanding of effective neurorehabilitation techniques, contributing to the fields of occupational therapy and physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Diagnoses of established stroke
* Present limitations or motor response deficiencies in the upper limb
* Maintain cognitive functions with the ability to follow the instructions of the interventions and evaluations (MOCA>14)

Exclusion Criteria:

* Diagnosed with mental illness before the stroke
* Other systemic conditions on the central nervous system
* Cardiorespiratory system pathologies in severe cases
* Acute period, fever, muscle inflammation or myopathies
* Any type of vascular and organic insufficiency
* Liver disease or skin lesions in the area of application of the electrodes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Data collection forms include gender identity questions, and the gender identity is sellf-determined by participants
Enrollment: 28 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Disability and Dependence Level - Barthel Index | Administered once, typically taking a few minutes.
  A general measure assessing patient independence, evaluating performance in basic daily activities (ADLs).
Upper Limb Functionality - Action Research Arm Test (ARAT) | Administration time ranges from 5 to 15 minutes.
  Assesses upper limb functionality post-cortical injury, involving manipulation tasks with various objects.
Cognitive Impairment - Montreal Cognitive Assessment (MoCA) | takes about 10 minutes for administration.
  Evaluates mild cognitive dysfunctions across multiple domains, including attention, memory, language, and executive functions.
Perception Impairment - Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | Duration varies based on the number and type of subtests administered.
  Specific for occupational therapy in stroke patients, assessing visual, spatial, motor, and cognitive perception.
Mental Evocation Ability - Mental Evocation of Images, Movements, and Activities Questionnaire (CEMIMA) | Duration varies
  Measures the ability to mentally form visual and kinesthetic images of the hand/upper limb.
Quality of Life Perception - Stroke Impact Scale 16 (SIS-16) | 5-10 minutes.
  A self-report measure focusing on physical aspects including strength, hand function, mobility, and ADLs.
Electromyographic Activity During MI and AO | during the experimental setup
  muscle activity using surface electrodes on wrist extensors and flexors.

SECONDARY OUTCOMES:
Age | 1 minute
  birth age
gender | 1 minute
  he gender with which the participant identifies
Marital Status | 1 minute
  single, married, divorced
Education Level | 1 minute
  he highest level of education
Economic Status | 1 minute
  participant's economic
Affected Side | 1 minute
  The side of the body affected by the stroke or injury
Dominant Side | 1 minute
  The side of the body that is the participant's natural dominant side
Type of Lesion | 1 minute
  specific type of brain injury
Time Since Injury | 1 minute
  time since the participant had the brain injury or stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salmanca, Salamanca, Salamanca, Spain